CLINICAL TRIAL: NCT05092672
Title: Impact of Traffic-related Air Pollution on the Cardiovascular and Pulmonary Response to Physical Activity in Patients With Hypertension
Brief Title: Physical Activity, Air Pollution, and High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Koehle, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H21-01487
Record Dates: First submitted 2021-09-28; First posted 2021-10-25 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Essential Hypertension
Keywords: Traffic-related air pollution; Physical activity; Exercise; Blood pressure; Heart rate variability; Arterial stiffness; Microvascular responsiveness; Muscle oxygen saturation; Lung function
MeSH Terms: conditions — Essential Hypertension; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High traffic-related air pollution first (Experimental): Participants will exercise in an environment with high levels of traffic-related air pollution first. Afterwards, participants will complete the same exercise in an environment with low levels of traffic-related air pollution.
  Interventions: Behavioral: Exercise
- Low traffic-related air pollution (Experimental): Participants will exercise in an environment with low levels of traffic-related air pollution first. Afterwards, participants will complete the same exercise in an environment with high levels of traffic-related air pollution.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will engage in moderate-intensity (40-59% HRR) exercise for 30 min

SUMMARY:
The investigators are investigating the effects of traffic-related air pollution (TRAP) on the cardiovascular and pulmonary response to exercise in patients with hypertension using a real world randomized, crossover study design. Participants will be exposed to 2 conditions: a low TRAP environment and a high TRAP environment. Each exposure will consist of 30 min of moderate-intensity exercise. Cardiovascular and pulmonary health outcomes will be measured before, during, and up to 24 hours following exposures. A minimum washout period of 1 week will be used to minimize carryover effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-70 years of age
2. Previously diagnosed with elevated blood pressure or hypertension by a physician

Exclusion Criteria:

1. Current or ex-smokers (abstinent for less than one year)
2. Lives with an individual who currently smokes cigarettes, e-cigarettes (i.e., vaping), or cannabis
3. Hormone replacement therapy use
4. Currently on beta-blocker or angiotensin receptor blocker (ARB) therapy
5. Currently using over the counter drugs or supplements that may alter cardiovascular measures (as per the principal investigator's discretion)
6. Prior diagnosis of any other existing cardiovascular or pulmonary diseases and/or conditions (other than hypertension)
7. Musculoskeletal injury or lower limb limitation preventing safe engagement in moderate-intensity exercise

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Blood Pressure at 2 Hours Post-Exposure | Baseline and 2 hours post-exposure
  MAP, SBP, and DBP

SECONDARY OUTCOMES:
24-Hour Blood Pressure | 24 hours post-exposure
  MAP, SBP, and DBP
Heart Rate Variability | Baseline and up to 24 hours post-exposure
  Indices of heart rate variability
Change from Baseline Arterial Stiffness at 2 Hours Post-Exposure | Baseline and 2 hours post-exposure
  Pulse wave velocity and augmentation index
Change from Baseline Microvascular Responsiveness at 2 Hours Post-Exposure | Baseline and 2 hours post-exposure
  Microvascular responsiveness (measured by near-infrared spectroscopy)
Muscle Oxygen Saturation | Continuously throughout the 30 minute exercise bouts (during exposure)
  Muscle oxygen saturation (measured by near-infrared spectroscopy)
Change from Baseline FEV1 and FVC at 2 Hours Post-Exposure | Baseline and 2 hours post-exposure
  Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) measured by spirometry (in L)
Change from Baseline FEV1/FVC at 2 Hours Post-Exposure | Baseline and 2 hours post-exposure
  FEV1/FVC ratio measured by spirometry
Change from Baseline FEF25-75 and PEFR at 2 Hours Post-Exposure | Baseline and 2 hours post-exposure
  Forced expiratory flow at 25-75% of forced vital capacity (FEF25-75) and peak expiratory flow rate (PEFR) measured by spirometry (in L/s)
Severity of Symptoms | Baseline and 2 hours post-exposure
  Severity of respiratory symptoms (e.g., dyspnea, cough, wheeze, chest tightness) and headache on a 0-5 scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koehle, MD, PhD, Principal Investigator — Professor
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No